CLINICAL TRIAL: NCT07160855
Title: Comparison of Letrozole With Misoprostol Versus Misoprostol Alone in the Management of Missed Miscarriages
Brief Title: Letrozole Plus Misoprostol Versus Misoprostol Alone for Treating Women With Missed Miscarriage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Afrayshum Tariq, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1327-5077
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Miscarriage in First Trimester; Missed Miscarriage
Keywords: Abortion, missed; Abortion, induced; Letrozole; Misoprostol; first trimester
MeSH Terms: conditions — Abortion, Incomplete; Abortion, Missed | interventions — Misoprostol; Arthrotec; Letrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol with placebo (Active Comparator): Vaginal Misoprostol will be instituted after oral placebo
  Interventions: Drug: Misoprostol (given vaginally); Drug: Placebo
- Misoprostol with Letrozole (Experimental): After oral letrozole, vaginal Misoprostol will be instituted
  Interventions: Drug: Misoprostol (given vaginally); Drug: Letrozole 5 mg

INTERVENTIONS:
Drug: Misoprostol (given vaginally) — 800 micrograms of a single dose of vaginal misoprostol will be given
  Other Names: Cytotec; Arthrotec
Drug: Letrozole 5 mg — 10 mg oral letrozole for 3 days will be given
  Other Names: femara
  Arms: Misoprostol with Letrozole
Drug: Placebo — oral placebo for three days will be given
  Arms: Misoprostol with placebo

SUMMARY:
The goal of this clinical trial is to learn whether adding the medicine letrozole to Misoprostol helps women have a complete abortion more often than using Misoprostol alone for the treatment of missed miscarriage (when a pregnancy has stopped developing but has not yet passed naturally).

The main questions this study aims to answer are:

1. Does taking letrozole for 3 days before misoprostol increase the chance of a complete abortion compared to misoprostol alone?
2. Does the use of letrozole affect the time it takes for abortion to occur? Who can Join? i. Women up to 13 weeks of pregnancy (based on last menstrual period and confirmed by ultrasound) who have a missed miscarriage.

ii. Only those with a single pregnancy are eligible. iii. Women with a previous cesarean section or uterine scar are not included.

What Will Happen in the Study A total of 92 women will take part.

Participants will be randomly assigned to one of two groups:

Group A: Letrozole tablets once daily for 3 days, followed by one dose of vaginal misoprostol.

Group B: Placebo tablets for maximum of 3 days, followed by one dose of vaginal misoprostol.

Doctors will monitor whether the abortion is complete within 24 hours. If it is not, other medical procedures will be offered as needed.

Products of conception will be examined to confirm abortion.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women up till 13th weeks of gestation according to last menstrual period (LMP) dates, confirmed on ultrasound
* Single intrauterine pregnancy
* Planned for termination due to missed miscarriage

Exclusion Criteria:

* Previous history of cesarean section
* Uterine scar due to previous procedure like myomectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Complete abortion | From start of study medication after randomization to within 24-hours
  The expulsion of both fetus and placenta without operative intervention and no retained products of conception confirmed on ultrasound.

OTHER OUTCOMES:
Induction-abortion interval | From start of study medication to abortion, within 24-hours
  The time interval (in hours) from the administration of first dose of Misoprostol up to the time when the fetus aborted.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia R Assistant Professor, FCPS, Study Chair — Nishtar Medical University and Hospital
Locations (1):
- Nishtar Medical University and Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasalizadeh F, Sahhaf F, Sadeghi-Shabestari P, Mirza-Aghazadeh-Attari M, Naghavi-Behzad M. Comparison Between Effect of Letrozole Plus Misoprostol and Misoprostol Alone in Terminating Non-Viable First Trimester Pregnancies: A Single Blind Randomized Trial. J Family Reprod Health. 2018 Mar;12(1):27-33. PMID 30647756